CLINICAL TRIAL: NCT03313596
Title: Multicenter Randomized Controlled Trial of Adenovirus-mediated Adjuvant Gene Therapy Improving Outcome of Liver Transplantation in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Multicenter RCT of ADV-TK Gene Therapy Improving the Outcome of Liver Transplantation for Advanced HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Beijing YouAn Hospital (Other)
Responsible Party: Principal Investigator, Ding Ma, Director, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LT-03
Record Dates: First submitted 2017-10-08; First posted 2017-10-18 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LT-only (Active Comparator): patients received orthotopic LT and subsequent immunosuppression therapy
  Interventions: Procedure: LT
- LT+ADV-TK (Experimental): ADV-TK therapy was administered in addition to orthotopic LT and subsequent immunosuppression therapy
  Interventions: Drug: ADV-Tk; Procedure: LT

INTERVENTIONS:
Drug: ADV-Tk — The first ADV-TK dose was administered during the operation; 1.0×10(12) viral particles of ADV-TK in 100 mL of 0.9% saline were injected into peritoneum tissues around the liver. The second and third ADV-TK dose was administered 60 days and 90 days after LT; 1.0×10(12) viral particles of ADV-TK in 100 mL of 0.9% saline were injected into the celiac artery (60 mL) and the superior mesenteric artery (40 mL) via femoral-artery puncture.
  Arms: LT+ADV-TK
Procedure: LT — Orthotopic LT and subsequent immunosuppression therapy

SUMMARY:
Compare the effect of liver transplantation (LT) plus ADV-TK gene therapy versus LT only in advanced primary hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years of age (Male and Female).
* Clinical diagnosis of advanced primary hepatocellular carcinoma who could accept liver transplantation.
* Patients who had unresectable HCC with single tumor diameter > 5 cm and ≤ 10cm; or numbers of multiple tumors >3 and ≤ 5, and the total length of foci diameter ≤ 15 cm.
* Serum AFP ≤ 10000 ng/ml before liver transplantation.
* Child-pugh A-B.
* No metastasis in extrahepatic main vescular and extrahepatic lymph node detected during the operation and no metastasis of other organs.
* Provide written informed consent before screening.

Exclusion Criteria:

* Metastasis in extrahepatic organs.
* HCC with Invasion in extrahepatic main vescular and extrahepatic organs.
* Contraindications of operation of other organ system.
* Hypersensitivity to adenovirus, GCV or similar drugs.
* Serious obstacle of the mechanism of coagulation, hemorrhagic tendency, and abnormal coagulation (≥50%).
* Plan to accept clinical trials of other antitumor drugs.
* Immunological deficit.
* HBsAg(+) and HBcAb(+) donor.
* Unsuitable participate assessed by investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2013-03; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival, PFS | 2-year
  PFS was measured from the day of liver transplantation to objective recurrence (MRI or CT) or HCC-related death, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival, OS | 1-year
  OS was measured from the day of liver transplantation to death.
Overall survival, OS | 2-year
  OS was measured from the day of liver transplantation to death.
Time of the tumor progression,TTP | 2-year
  TTP was the median period from the day of liver transplantation to objective recurrence (MRI or CT).
Median overall survival time | 2-year

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Beijing Youan Hospital, Beijing, Beijing Municipality
  - 301 Military Hospital, Beijing
  - General Hospital of Chinese People's Armed Police, Beijing
  - The Third XiangYa Hospital of Central South University, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - The Third Affiliated Hospital,Sun Yat-sen University, Guangzhou
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - Zhongshan Hospital of Fudan University, Shanghai
  - The First Affiliated Hospital of China Medical University, Shenyang
  - The First Center Hospital of Tianjin, Tianjin
  - The First Hospital of Xinjiang Medical University, Ürümqi